CLINICAL TRIAL: NCT03873363
Title: Prospective Randomized Comparison of Cruciate-retaining and Cruciate Substituting Surgical Technique for Total Knee Arthroplasty
Brief Title: Clinical Outcome After Total Knee Arthroplasty Using CR or PS Inlay
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TKA CR vs PS
Record Dates: First submitted 2019-03-07; First posted 2019-03-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Arthroplasty; Total Knee Replacement; Outcome; Implant Design
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomization to one of two surgical techniques.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PS (Experimental): Implantation of a posterior stabilized (cruciate substituting) Total Knee Arthroplasty.
  Interventions: Device: PS TKA
- CR (Active Comparator): Implantation of a cruciate retaining Total Knee Arthroplasty.
  Interventions: Device: CR TKA

INTERVENTIONS:
Device: PS TKA — Implantation of a posterior stabilized (cruciate substituting) Total Knee Arthroplasty.
  Arms: PS
Device: CR TKA — Implantation of a cruciate retaining Total Knee Arthroplasty.
  Arms: CR

SUMMARY:
Compare knee flexion after cruciate-retaining and cruciate substituting Total Knee Arthroplasty.

DETAILED DESCRIPTION:
The aim of this study is to compare knee Flexion after cruciate-retaining (CR) and cruciate-substituting (posterior stabilized - PS) Total Knee Arthroplasty (TKA).

For this purpose, flexion and extension of the knee joint are measured using a goniometer preoperatively and up to ten years after surgery In addition, the clinical outcome will be assessed and evaluated using internationally recognised and evaluated scores (Knee Society Score, Oxford Knee Score, EQ5D, UCLA Activity Score).

Patients are randomized to receive a PS or CR TKA. Patients are assessed before surgery, after 3 months, 1 year, 2 years, 5 years, 7 years and 10 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Indication for TKA with a non-linked, bicondylar total knee replacement
* written informed consent

Exclusion Criteria:

* Chronic pain patients
* Neuromuscular Diseases
* general illnesses that make mobilisation more difficult and/or prevent follow-up
* Known posterior cruciate ligament insufficiency
* Need for a higher degree of linkage
* BMI over 40 kg/m²
* Study doctor, his family, employees or other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Knee Flexion | 1 year after surgery
  Knee flexion measured using a goniometer

SECONDARY OUTCOMES:
Function assessed by the Knee Society Score | 10 years after surgery
  Knee Society Score
Patient Reported Outcome | 10 years after surgery
  Oxford Knee Score
Health-related Quality of Life | 10 years after surgery
  EQ-5D-3L
Activity assessed by UCLA activity score | 10 years after surgery
  UCLA activity score

OTHER OUTCOMES:
Adverse Events | 1 year after surgery
  Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- University Center of Orthopaedics and Traumatology, University Medicine Carl Gustav Carus Dresden, TU Dresden, Dresden, Saxony, Germany